CLINICAL TRIAL: NCT03168269
Title: Can CCTA Technicians Provide Accurate Interpretation of Findings in Chest Pain Patients Presenting to the Emergency Department in After Hours?
Brief Title: Can CCTA Technicians Provide Accurate Interpretation of Findings in Patients Presenting to the ED in After Hours?
Status: Completed | Type: Observational
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Sponsor
Other Study IDs: JorCCTA
Record Dates: First submitted 2017-04-29; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Coronary Artery Disease
Keywords: CCTA interpretation; technicians; experts; comparison
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Coronary Computed Tomographic Angiography (CCTA) — CCTA of coronary arteries

SUMMARY:
Coronary Computed Tomographic Angiography (CCTA) is emerging as the diagnostic test of choice in chest pain patients with low to intermediate probability of coronary artery disease (CAD). Qualified CCTA readers may not be available around the clock in most centers, limiting the use of CCTA. This study aimed to determine if well-qualified CCTA technicians can provide initial accurate diagnosis to guide initial management and triage of such patients

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for elective CCTA to assess coronary artery disease

Exclusion Criteria:

* Patients with previous coronary revascularization procedures (PCI or CABG).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients referred from the ED or outpatient service for elective CCTA to rule out CAD
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2016-02-25 (Actual); Study Completion 2016-02-25 (Actual)

PRIMARY OUTCOMES:
The agreements between the two technicians and the cardiologist in evaluation of coronary segments | 24 hours
  All coronary segments are independently assesses for CAD by the two technicians and the expert cardiologist

IPD SHARING:
Plan to Share IPD: Undecided